CLINICAL TRIAL: NCT03250130
Title: Medical Ericksonian Hypnosis on Patients Treated With Adjuvant Chemotherapy for Breast Cancer at the ICM Val d'Aurelle - Montpellier: a Feasibility Study
Brief Title: Hypnosis for Patients Treated With Adjuvant Chemotherapy for Breast Cancer(HYPNOVAL)
Acronym: HYPNOVAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut du Cancer de Montpellier - Val d'Aurelle (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: ICM-URC-2014/ 31
Record Dates: First submitted 2016-08-29; First posted 2017-08-15 (Actual); Last update posted 2020-08-10 (Actual); Status verified 2020-08

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Hypnosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Hypnosis (Experimental): The patient achieve self-hypnosis sessions in these chemotherapy treatments
  Interventions: Behavioral: hypnosis

INTERVENTIONS:
Behavioral: hypnosis — The patient achieve self-hypnosis sessions in these chemotherapy treatments

SUMMARY:
The main objective is to assess the feasibility of an intervention based on medical Ericksonian hypnosis as a complementary therapy in patients treated with surgery after a diagnosis of breast cancer, followed by an indication of adjuvant chemotherapy and radiotherapy

DETAILED DESCRIPTION:
In the field of management of cancer, many approaches have been used since tens of years, particularly in regard of pain management, both in achieving surgical or invasive procedures in the pain induced by the disease itself. the investigators owe the first description in 1829 Chapelin and col who used hypnosis in a patient with breast cancer in which a mastectomy should be performed. Meta-analysis (2000) showed the positive impact of analgesia obtained through hypnosis on the perception of pain intensity. In children in whom regular venous punctures is performed, using hypnosis seems indisputable on the management of anticipatory anxiety, leading to a better experience of the act itself. Regarding the nausea and vomiting induced by chemotherapy, numerous studies are old, not always randomized and performed often before the era of the setrons; but seems favorable impact on anticipated nausea and vomiting, the updated studies should emerge on the issue of delayed emesis which remain a serious adverse event and not completely resolved. Mark to improve the EORTC validated tools of quality of life measurement widely used for example in ovarian cancer.

The impact of hypnosis on the quality of life or the side effects of treatment or rehospitalization for toxicity remains controversial (Judson, 2011). A meta-analysis combining the tests carried out before and after the era of setrons (Richardson, 2007) concluded that the effectiveness of the anticipated nausea and vomiting.

In this context,the investigators proposed to conduct a feasibility study to evaluate the role and impact of medical Ericksonian hypnosis on acute and delayed adverse event (incl nausea and vomiting) in female patients treated by adjuvant chemotherapy for breast cancer.

The main objective is to assess the feasibility of an intervention based on medical Ericksonian hypnosis as a complementary therapy in patients treated with surgery after a diagnosis of breast cancer, followed by an indication of adjuvant chemotherapy and radiotherapy

ELIGIBILITY:
Inclusion Criteria:

* • Female, age > 18 years-old

  * Without previous practice of hypnosis
  * Patient with diagnosis of breast cancer
  * Patient receiving an adjuvant chemotherapy for at least 3 months with an indication of radiotherapy after chemotherapy
  * Patient accepting the principle of the study with a signed written informed consent
  * Patient affiliated to French Social Security

Exclusion Criteria:

* • Male

  * Age < 18 years
  * Patient refusing hypnosis
  * Pregnancy, breast-feeding, or lack of effective contraception in female patients with reproductive potential.
  * Patient with psychological or mental disorders under psychotropic treatments (lithium, neuroleptics)
  * Not ability to speak and read French, deaf and/or mute

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2015-07-01 (Actual); Primary Completion 2016-09-01 (Actual); Study Completion 2017-06-06 (Actual)

PRIMARY OUTCOMES:
proportion of patients rated as being compliant to self-hypnosis | through study completion, an average of 2 years
  The main objective is to assess the feasibility of an intervention based on medical Ericksonian hypnosis as a complementary therapy in patients treated with surgery after a diagnosis of breast cancer, followed by an indication of adjuvant chemotherapy and radiotherapy.
  Primary endpoint is the proportion of patients rated as being compliant to self-hypnosis sessions during adjuvant chemotherapy (6 sessions). A patient is considered as compliant if it achieves at least 2/3 of the planned self-hypnosis sessions, that is, 4 of 6 planned sessions.

SECONDARY OUTCOMES:
Impact of hypnosis on the tolerance of the CT | through study completion, an average of 2 years
  The secondary objective is to describe its impact on the tolerance of the CT

CONTACTS AND LOCATIONS:
Overall Officials: Michel FABBRO, Study Chair — Institut régional du Cancer de Montpellier
Locations (1):
- Institut régional du Cancer de montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: No